CLINICAL TRIAL: NCT02465151
Title: Assessment of the Optimal Amount of Proteins at Breakfast for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14.09.NRC
Record Dates: First submitted 2015-05-21; First posted 2015-06-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Children

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Protein (Experimental)
  Interventions: Other: Protein-based beverage
- Low Protein (Experimental)
  Interventions: Other: Protein-based beverage
- Medium Protein (Experimental)
  Interventions: Other: Protein-based beverage
- High Protein (Experimental)
  Interventions: Other: Protein-based beverage

INTERVENTIONS:
Other: Protein-based beverage — protein-based beverage

SUMMARY:
The primary objective of this trial is to identify how much protein is required at breakfast to promote positive whole body protein balance over the following 9h period.

DETAILED DESCRIPTION:
This study will be the first to establish the role of eating protein at breakfast on whole body protein balance in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7-12 years of age
* Healthy and recreationally physically active (obtaining a 3- day average moderate/vigorous physical activity of at least 30 min/day)
* Body mass at ≥10th percentile for 7 year olds and ≤85th percentile for 12 year olds. Values based upon 2000 CDC Growth Charts for the United States
* Having obtained his/her informed assent
* Having obtained his/her consent from parent or legal guardian
* Being able to communicate in local language
* Have a habitual daily protein consumption of between 1.6 g/kg and 2.4 g/kg/bw

Exclusion Criteria:

* Self-report on regular medication impacting the metabolism, such as corticoids, hormone (e.g thyroid, adrenal) treatment, or medication against diabetes or against hypercholesterolemia or hypertriglyceridemia
* Self-reported history of metabolic, hepatic or renal disease
* Self-reported allergy to milk proteins (e.g., whey or casein) or intolerance to any food ingredients to be used in the study products and meals
* Within 1.5 years of estimated age of peak height velocity (PHV)
* Special diet or weight loss program (e.g Atkins diet)
* Consuming breakfast containing more than 21g of protein on each day of the 3-d screening period
* Subject who cannot be expected to comply with the study procedures, including unwillingness to consume study product and meals
* Currently participating or having participated in another nutritional-clinical trial during the last 2 months prior to the beginning of this study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Whole body protein balance (g protein/9 hours) by nitrogen balance technique | 9 hours following ingestion of investigational product

SECONDARY OUTCOMES:
Whole body protein balance (g protein/24 hours) by nitrogen balance technique | 24 hours following ingestion of investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Dan Moore, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport at University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karagounis LG, Volterman KA, Breuille D, Offord EA, Emady-Azar S, Moore DR. Protein Intake at Breakfast Promotes a Positive Whole-Body Protein Balance in a Dose-Response Manner in Healthy Children: A Randomized Trial. J Nutr. 2018 May 1;148(5):729-737. doi: 10.1093/jn/nxy026. PMID 30053279